CLINICAL TRIAL: NCT00964730
Title: A Phase I, Single-Center, Double-Blind, Randomized, Placebo- and Positive- Controlled, Parallel Group, Thorough QT/QTc Study to Evaluate the Effect of Talampanel on Cardiac Repolarization in Healthy Male and Female Volunteers
Brief Title: A Phase 1 Study to Investigate the Effects of Talampanel on the Heart Rhythm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Siyu Liu, M.D., Ph.D. VP, Teva Neuroscience, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAL-TQT-101; R09-0539
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Thorough QT Study; Talampanel; Cardiac Repolarizatiom; Healthy Volunteers
MeSH Terms: interventions — talampanel; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Talampanel (Experimental)
  Interventions: Drug: Talampanel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Other)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Talampanel — titrated to 50mg three times a day over 9 days and a single dose administered on Day 10
  Other Names: TV-7600, GYKI 53773
  Arms: Talampanel
Drug: Moxifloxacin — Placebo administered three times a day over 9 days and a single dose of moxifloxacin administered on Day 10
  Other Names: Avelox
  Arms: Moxifloxacin
Drug: Placebo — administered three times a day over 9 days and a single dose administered on Day 10
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether multiple doses of Talampanel increase the QT interval when compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 50 years of age inclusive.
* Body mass index: Between 18 and 30 kg/m2 and weight of at least 50 kg.
* Female volunteers must have either a negative pregnancy test and be willing to use birth control, be post-menopausal evidenced by lab test, or be surgically sterile.
* Volunteers must be able to understand the requirements of the study and must be willing to comply with the requirements of the study and provide their written informed consents to participate in the study prior to the conduct of study procedures.

Exclusion Criteria:

* Male and female volunteers with a resting QT interval of < 320 msec or > 450 msec (males) or > 470 msec (females
* Volunteers with ECG abnormalities that may interfere with the accurate assessment of the QT interval
* Volunteers with known cardiovascular disorders, including coronary artery disease, valvular heart disease, cardiomyopathies, or ECG abnormalities suggestive of prior myocardial infarction, chamber enlargement or hypertrophy.
* Volunteers with known clinically significant arrhythmias or rhythm disturbances observed on ECG
* Volunteers who have a history of, or risk factors for, Torsades de Pointes (e.g. heart failure, abnormal serum electrolytes), including a history of family history of arrhythmia, sudden death, long QT syndrome, Brugada complex, or personal history of syncope.
* Volunteers who have a heart rate outside 40-90 beats per minute
* Volunteers who have a blood pressure outside 90-140 mmHg systolic or 45-90 mmHg diastolic
* Volunteers with history of uncontrolled hypertension, impaired glucose tolerance, diabetes mellitus, kidney disease, edema, stroke or neurological disorder, rheumatological disorder, lung disease, heart disease, liver disease, or a history of any illness that pose additional risk to the volunteer
* Volunteers with a history of psychiatric disorders, including bipolar disorder, psychosis, previous episode(s) of major depression, history of suicidality or suicidal ideation.
* Volunteers who have history of surgeries or conditions that affect the way drugs are absorbed or distributed in the body such as intestinal surgery, stomach surgery.
* Volunteers with impaired liver function and elevated liver enzymes
* Volunteers with major trauma or surgery in the past 2 months, acute infection within 2 weeks, cancer within the last 5 years (excluding non-melanoma skin cancers), History of tuberculosis, abnormal lab tests
* Female volunteers who are lactating or intend to become pregnant during the study period.
* Volunteers with a known allergy or sensitivity to moxifloxacin or its derivatives, benzodiazepines, talampanel or its derivatives, or any contraindications to moxifloxacin, benzodiazepines, or talampanel.
* Volunteers with significant food or drug allergies
* Volunteers that have used an investigational drug (new chemical entity) 3 months prior to the start of the study,.who have consumed any medications (including over-the-counter medications, prescription medications, investigational drugs, vitamins, or herbal remedies) within 30 days prior to check-in (with the exception of hormonal contraceptives [females only] and occasional use of acetaminophen and ibuprofens, who have consumed amiodarone and chloroquine within 4 months prior to screening, who have consumed excessive amounts of alcohol or are unwilling to comply with the restricted use of alcohol during the study, who have consumed excessive amounts of coffee, tea, coke, or other caffeinated beverages within 2 weeks prior to check-in, who have consumed quinine (tonic water) within 7 days prior to study start, who have consumed grapefruit, grapefruit juice, or Seville orange juice within the 7 days prior to study start, who smoke, have smoked in the last 3 months, or are planning to start smoking during the study, tobacco users, subjects currently using nicotine products, or subjects with a positive urine cotinine test at study start
* Volunteers who are currently regular users (including recreational use) of any illicit drugs or who have a history of drug (including alcohol) abuse within 1 year of study start.
* Volunteers with positive urine test for drugs of abuse at screening or check-in.
* Volunteers who have donated or received any blood, plasma, or platelet transfusions in the 3 months prior to study start, or who have made donations on more than two occasions within the 12 months preceding the first dose administration, or who have planned donations during the study or during the 3 months following the study.
* Volunteers with a positive screening test for Hepatitis B, Hepatitis C or HIV
* Volunteers not willing to refrain from changing level of activity during the study and from jogging and strenuous exercise of all types while at the research unit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine the effects of Talampanel on cardiac repolarization after multiple therapeutic doses administered over 10 days | 12 days

SECONDARY OUTCOMES:
Examine the PK profile of talampanel and its metabolite -Assess the PK/PD relationship of the time course of QT/QTc interval prolongation-Assess the safety and tolerability of multiple doses of talampanel in healthy volunteers | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Sprenger, MD, Principal Investigator — Cetero Research - Fargo
Locations (1):
- Cetero Research - Fargo, Fargo, North Dakota, United States